CLINICAL TRIAL: NCT01209832
Title: The Effect of Tasisulam on CYP3A-mediated Metabolism of Midazolam: A Pharmacokinetic Interaction Study in Cancer Patients With Advanced and/or Metastatic Tumors or Lymphoma
Brief Title: A Tasisulam and Midazolam Drug Interaction Study in Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated based on safety results from another trial
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13074; H8K-MC-JZAP (Other: Eli Lilly and Company); 2010-020090-16 (EudraCT Number)
Record Dates: First submitted 2010-09-23; First posted 2010-09-27 (Estimated); Results first posted 2019-03-18 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2018-12

CONDITIONS: Advanced Cancer
Keywords: Metastatic Tumors; Lymphoma
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoma | interventions — N-((5-bromo-2-thienyl)sulfonyl)-2,4-dichlorobenzamide; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug Interaction arm (Experimental)
  Interventions: Drug: Tasisulam; Drug: Midazolam

INTERVENTIONS:
Drug: Tasisulam — Patient specific dose, administered intravenously, on Day 1 of a 28-day cycle. Minimum of one (1) 28-day cycle. Patients may continue to receive tasisulam until disease progression or until discontinuation criteria are met.
  Other Names: LY573636
Drug: Midazolam — 1.2 milligrams (mg), administered orally once prior to the initiation of tasisulam therapy and once on Day 8 after initiation of tasisulam therapy

SUMMARY:
The purpose of this study is to evaluate whether tasisulam acts as an inducer of CYP3A using midazolam as a sensitive and specific probe substrate of CYP3A.

The study will also assess the safety and tolerability of tasisulam and midazolam given in combination and document any antitumor activity with tasisulam.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed solid malignancy or lymphoma that is advanced and/or metastatic disease which has not responded to standard therapy or for which no standard therapy exists.
* Have a performance status of less than or equal to 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, cancer-related hormonal therapy, or other investigational therapy for at least 30 days (45 days for mitomycin-C or nitrosoureas) prior to study enrollment and recovered from the acute effects of therapy. Limited field radiotherapy is permitted (in consultation with the investigator)
* Have an estimated life expectancy, in the judgment of the investigator, of greater than or equal to 12 weeks

Exclusion Criteria:

* Have received treatment within 30 days of the initial dose of study drug with an experimental agent for non-cancer indications that has not received regulatory approval for any indication
* Have symptomatic central nervous system (CNS) malignancy or metastasis (screening not required). Patients with active brain metastasis are excluded
* Have current acute or chronic leukemia
* Patients who have clinically significant chronic obstructive pulmonary disease (COPD) or other respiratory diseases that may be at risk during periods of conscious sedation under midazolam
* Patients with a known history of obstructive sleep apnea, difficult intubation, or syndromes associated with airway abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- France (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bordeaux
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes

RESULTS

PARTICIPANT FLOW:
Groups:
- Midazolam + Tasisulam: Period 1 (7 days): 1.2 milligrams (mg) midazolam orally on Day 1.
  Period 2 (28 days): Tasisulam intravenously to target area under the curve above the albumin corrected threshold (AUCalb) in the range of 1200 to 6400 hour*micrograms per milliliter (h*mcg/mL) on Day 1 and 1.2 mg midazolam orally on Day 8.
  Maintenance Period 1 and 2 (35 days): Tasisulam was dosed intravenously to target AUCalb in the range of 1200 to 6400 h*mcg/mL on Day 1.
Period: Period 1
Arm/Group | Midazolam + Tasisulam
Started | 11
Received At Least 1 Dose of Study Drug | 10
Completed | 10
Not Completed | 1
Not completed — Sponsor Decision and was not dosed | 1
Period: Period 2
Arm/Group | Midazolam + Tasisulam
Started | 10
Completed | 9
Not Completed | 1
Not completed — Sponsor Decision | 1
Period: Maintenance Period 1 (M1)
Arm/Group | Midazolam + Tasisulam
Started | 4 (Five participants who completed Period 2 did not enroll into Maintenance Period.)
Completed | 4
Not Completed | 0
Period: Maintenance Period 2 (M1)
Arm/Group | Midazolam + Tasisulam
Started | 3 (One participant who completed maintenance period 1 did not enter maintenance period 2.)
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug.
Groups:
- Midazolam + Tasisulam: Period 1 (7 days): 1.2 milligrams (mg) midazolam orally on Day 1.
  Period 2 (28 days): Tasisulam intravenously to target area under the curve above the albumin corrected threshold (AUCalb) in the range of 1200 to 6400 hour*micrograms per milliliter (h*mcg/mL) on Day 1 and 1.2 mg midazolam orally on Day 8.
  Maintenance Period (35 days): Tasisulam was dosed intravenously to target AUCalb in the range of 1200 to 6400 h*mcg/mL on Day 1.
Arm/Group | Midazolam + Tasisulam
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  France | 10

OUTCOME MEASURES:

1. Primary Outcome: Midazolam Pharmacokinetics: Area Under the Concentration-Time Curve From Time Zero to the Last Time Point With Measurable Concentrations (AUC 0-tlast)
Time Frame: Period 1 and 2: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 9, 11, 24, 48, and 72 hours post-dose.
Population: All participants who received study drug and had sufficient pharmacokinetics data to calculate AUC0-tlast. Analysis used data according to the treatment the participants actually received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Groups:
- Midazolam: Period 1 (7 days): 1.2 milligrams (mg) midazolam orally on Day 1.
- Midazolam + Tasisulam: Period 2 (28 days): Tasisulam was dosed intravenously to target area under the curve above the albumin corrected threshold (AUCalb) in the range of 1200 to 6400 hour*micrograms per milliliter (h*mcg/mL) on Day 1 and followed by 1.2 mg midazolam orally on Day 8.
Arm/Group | Midazolam | Midazolam + Tasisulam
Number analyzed (Participants) | 10 | 9
nanograms*hour per milliliter (ng*h/mL) | 25.9 (35) | 22.5 (55)

2. Primary Outcome: Midazolam Pharmacokinetics: Maximum Concentration (Cmax)
Time Frame: Period 1 and 2: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 9, 11, 24, 48, and 72 hours post-dose.
Population: All participants who received study drug and had sufficient pharmacokinetics data to estimate Cmax. Analysis used data according to the treatment the participants actually received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Midazolam | Midazolam + Tasisulam
Number analyzed (Participants) | 10 | 9
nanograms per milliliter (ng/mL) | 9.07 (41) | 9.48 (51)

3. Primary Outcome: Midazolam Pharmacokinetics: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC 0-infinity)
Time Frame: Period 1 and 2: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 9, 11, 24, 48, and 72 hours post-dose.
Population: All participants who received study drug and had sufficient pharmacokinetics data to calculate AUC0-infinity. Analysis used data according to the treatment the participants actually received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | Midazolam | Midazolam + Tasisulam
Number analyzed (Participants) | 9 | 9
nanograms*hour per milliliter (ng*h/mL) | 27.0 (36) | 22.8 (54)

4. Secondary Outcome: Number of Participants With Tumor Response
Description: Number of participants with tumor response = number of participants with complete response (CR) + number of participants with partial response (PR), as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) guidelines. CR is disappearance of all target and non-target lesions; PR is ≥30% decrease in sum of longest diameter of target lesions.
Time Frame: Baseline to Day 15 of Maintenance Period up to 3 months
Population: All participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam + Tasisulam
Number analyzed (Participants) | 10
Participants | 0

5. Secondary Outcome: Tasisulam Pharmacokinetics: Maximum Concentration (Cmax)
Time Frame: Period 2: Predose, preinfusion start, 1, 1.75, 2 (post end of infusion), 2.5, 3, 4, 6, 8, 24, 48, 72, 120, 168, and 336 hours.
Population: All participants who received tasisulam and had pharmacokinetics data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Groups:
- Tasisulam: Period 2 (28 days): Tasisulam was dosed intravenously to target area under the curve above the albumin corrected threshold (AUCalb) in the range of 1200 to 6400 hour*micrograms per milliliter (h*mcg/mL) on Day 1 and followed by 1.2 milligrams (mg) midazolam orally on Day 8.
Arm/Group | Tasisulam
Number analyzed (Participants) | 9
micrograms per milliliter (mcg/mL) | 358 (17)

6. Secondary Outcome: Tasisulam Pharmacokinetics: Area Under the Concentration-Time Curve Above the Albumin Corrected Threshold (AUCalb)
Description: Tasisulam is highly bound to albumin. AUCalb is a surrogate measure of exposure to unbound (free) tasisulam.
Time Frame: as for outcome 5
Population: All participants who received tasisulam and had pharmacokinetics data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*micrograms/milliliter (h*mcg/mL)
Arm/Group | Tasisulam
Number analyzed (Participants) | 9
hour*micrograms/milliliter (h*mcg/mL) | 5840 (50)

ADVERSE EVENTS:
Groups:
- Tasisulam and Midazolam: Period 2 (28 days): Tasisulam intravenously to target area under the curve above the albumin corrected threshold (AUCalb) in the range of 1200 to 6400 hour*micrograms per milliliter (h*mcg/mL) on Day 1 and 1.2 mg midazolam orally on Day 8.
- Tasisulam (M1): Maintenance Period 1 (35 days): Tasisulam was dosed intravenously to target AUCalb in the range of 1200 to 6400 h*mcg/mL on Day 1.
- Tasisulam (M2): Maintenance Period 2 (35 days): Tasisulam was dosed intravenously to target AUCalb in the range of 1200 to 6400 h*mcg/mL on Day 1.
Arm/Group | Midazolam | Tasisulam and Midazolam | Tasisulam (M1) | Tasisulam (M2)
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 7/10 | 9/10 | 2/4 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam (N=10) | Tasisulam and Midazolam (N=10) | Tasisulam (M1) (N=4) | Tasisulam (M2) (N=3)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam (N=10) | Tasisulam and Midazolam (N=10) | Tasisulam (M1) (N=4) | Tasisulam (M2) (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days